CLINICAL TRIAL: NCT06471361
Title: A Multicenter, Open-Label, Outpatient Study to Evaluate the Safe And Effective Use of a Zilucoplan Auto-Injector Combination Product for Subcutaneous Self-Administration by Study Participants With Generalized Myasthenia Gravis
Brief Title: A Study to Evaluate the Safe and Effective Use of a Zilucoplan Auto-injector by Study Participants With Generalized Myasthenia Gravis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DV0013; U1111-1302-4369 (Other: World Health Organization (WHO)); 2023-508287-30 (Registry Identifier: EU Clinical Trials)
Record Dates: First submitted 2024-06-18; First posted 2024-06-24 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Generalized Myasthenia Gravis
Keywords: gMG
MeSH Terms: conditions — Myasthenia Gravis | interventions — zilucoplan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Zilucoplan-auto-injector (ZLP-AI) (Experimental): Study participants will self-administer zilucoplan (ZLP) based on their body weight using auto-injector (AI).
  Interventions: Drug: Zilucoplan

INTERVENTIONS:
Drug: Zilucoplan — Zilucoplan will be self-administered subcutaneously by study participants at pre-specified time points.
  Other Names: RA101495

SUMMARY:
The purpose of this study is to evaluate the effectiveness, safety and tolerability of zilucoplan auto-injector (ZLP-AI) self-administration.

ELIGIBILITY:
Inclusion Criteria:

* Study participant is male or female and must be at least 18 years of age at the time of signing the informed consent form (ICF).
* Study participant must have a documented diagnosis of gMG, based on study participant's history and supported by previous evaluations.
* Study participant is currently participating in ZLP (zilucoplan) study RA101495-02.302 (NCT04225871) or is administering commercial ZLP on a stable dosing regimen for at least 1 month prior to Screening.
* Study participants on commercial ZLP need to receive ZLP per the approved local labeling.
* Study participant is considered reliable and capable of adhering to the study protocol (eg, able to understand and complete questionnaires and able to adhere to the visit schedule) according to the judgement of the Investigator.
* Study participant is willing and capable of self-administering ZLP using the zilucoplan-auto-injector (ZLP AI) according to the instructions for use (IFU), ie, does not have any visual, physical, or other disability or impairment that interferes with his/her capacity to self-administer; if the participant has a caregiver, he/she may assist the participant with the injection.
* Vaccination with a quadrivalent meningococcal vaccine and, where available, meningococcal serotype B vaccine at least 14 days prior to investigational medicinal product (IMP) administration, if not vaccinated within 3 years prior to the start of treatment. Booster vaccination(s) should also be administered as clinically indicated, according to the local standard of care, for participants who have been previously vaccinated against Neisseria meningitidis.
* Female participants of childbearing potential must have a negative urine pregnancy test prior to the first dose of study drug.
* Male and/or female study participants

  1. A male participant must agree to use contraception during the Treatment Period and for 40 days after the last dose of study medication, and refrain from donating sperm during this period.
  2. A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least 1 of the following conditions applies:
* Not a woman of childbearing potential (WOCBP) OR A WOCBP who agrees to follow the contraceptive guidance the Treatment Period and for 40 days after the last dose of study medication.
* Capable of giving signed informed which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.

Exclusion Criteria:

* Study participant has any medical or psychiatric condition that, in the opinion of the Investigator, could jeopardize or would compromise the study participant's ability to participate in this study.
* Female participants who are breastfeeding, pregnant, or plan to become pregnant during the study.
* Study participant has a known hypersensitivity to any components of the study medication (and/or an investigational device) as stated in this protocol.
* Study participant has a clinically relevant active infection or a history of serious infection (resulting in hospitalization or requiring intravenous antibiotic treatment) within 6 weeks before Visit 1.
* Study participant has a history of meningococcal disease.
* Participant has previously participated in this study or participant has previously been assigned to treatment in a study of the medication under investigation in this study (except studies RA101495-02.201 (NCT03315130), RA101495-02.301 (NCT04115293), or RA101495-02.302 (NCT04225871), which are not excluded, unless the participant was required to withdraw from said studies for a safety reason which could reasonably recur).
* Participant has participated in another study of an IMP (and/or an investigational device) different from ZLP within the previous 3 months or 5 half-lives, whichever is longer, or is currently participating in another study of an IMP (and/or an investigational device).
* Current unstable liver or biliary disease at Screening (Visit 1), per Investigator assessment, defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, persistent jaundice, or cirrhosis. NOTE: with exception of stable hepatobiliary conditions (including Gilbert's syndrome, asymptomatic gallstones).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2024-08-27 (Actual); Primary Completion 2025-01-28 (Actual); Study Completion 2025-02-03 (Actual)

PRIMARY OUTCOMES:
Percentage of effective self-administrations of zilucoplan using the zilucoplan-auto-injector (ZLP-AI) from Visit 1 to Visit 8 | Visit 1 (Day 1) to Visit 8 (Day 14)
  Effective self-administration is defined as: Complete dose delivery: completeness of the delivery as confirmed by the Investigator. The entire dose of investigational medicinal product (IMP) should be completely delivered (that is, the yellow plunger that can be seen through the device window should be completely depressed).

SECONDARY OUTCOMES:
Percentage of effective self administrations of zilucoplan using ZLP-AI at Visit 8 | Visit 8 (Day 14)
  Effective self-administration is defined as: Complete dose delivery: completeness of the delivery as confirmed by the Investigator. The entire dose of IMP should be completely delivered (that is, the yellow plunger that can be seen through the device window should be completely depressed).
Percentage of effective self administration of zilucoplan using ZLP-AI at Visit 1 | Visit 1 (Day 1)
  Effective self-administration is defined as: Complete dose delivery: completeness of the delivery as confirmed by the Investigator. The entire dose of IMP should be completely delivered (that is, the yellow plunger that can be seen through the device window should be completely depressed).
Occurrence of serious adverse events (SAEs) during the course of the study | From Visit 1 (Day 1) up to the Safety Follow-up Visit (up to Day 21)
  A SAE is defined as any untoward medical occurrence that, at any dose: a. Results in death; b. Is life-threatening; c. Requires inpatient hospitalization or prolongation of existing hospitalization; d. Results in persistent disability/incapacity; e. Is a congenital anomaly/birth defect; f. Important medical events.
Occurrence of treatment-emergent adverse events (TEAEs) during the course of the study | From Visit 1 (Day 1) up to the Safety Follow-up Visit (up to Day 21)
  Treatment-emergent adverse events (TEAEs) are any untoward medical incidence in a subject during administered study treatment, whether or not these events are related to study treatment.
Occurrence of nonserious adverse device effects (ADE) during the course of the study | From Visit 1 (Day 1) up to the Safety Follow-up Visit (up to Day 21)
  An ADE is defined as an adverse event related to the use of an investigational medical device. This definition includes any adverse events resulting from insufficient or inadequate instructions for use, deployment, implantation, installation, or operation, or any malfunction of the investigational medical device as well as any event resulting from use error or from intentional misuse of the investigational medical device.
Occurrence of serious adverse device effects (SADE) during the course of the study | From Visit 1 (Day 1) up to the Safety Follow-up Visit (up to Day 21)
  A SADE is defined as an adverse device effect that has resulted in any of the consequences characteristic of a serious adverse event. A SAE is defined as any untoward medical occurrence that, at any dose: a. Results in death; b. Is life-threatening; c. Requires inpatient hospitalization or prolongation of existing hospitalization; d. Results in persistent disability/incapacity; e. Is a congenital anomaly/birth defect; f. Important medical events.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273
Locations (11):
- United States (7):
  - Dv0013 50628, New Haven, Connecticut
  - Dv0013 50634, Tampa, Florida
  - Dv0013 50648, Columbia, Missouri
  - Dv0013 50556, Chapel Hill, North Carolina
  - Dv0013 50635, Columbus, Ohio
  - Dv0013 50555, Austin, Texas
  - Dv0013 50636, Greenfield, Wisconsin
- Poland (3):
  - Dv0013 40609, Katowice
  - Dv0013 40759, Krakow
  - Dv0013 40605, Poznan
- Dv0013 40760, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed.All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: https://www.Vivli.org